CLINICAL TRIAL: NCT00121446
Title: Which Early ST Elevation Myocardial Infarction Therapy? The WEST Study
Brief Title: Which Therapy for Acute Heart Attacks? (The WEST Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry); Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVC1002
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2005-07

CONDITIONS: Myocardial Infarction
Keywords: Heart Attack; ST Elevation Myocardial Infarction; fibrinolytic therapy; percutaneous coronary intervention; Acute Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Tenecteplase; Enoxaparin; Clopidogrel; Percutaneous Coronary Intervention

INTERVENTIONS:
Drug: tenecteplase
Drug: enoxaparin
Drug: clopidogrel
Procedure: percutaneous coronary intervention

SUMMARY:
In the setting of acute myocardial infarction (heart attacks), the principle objective of the WEST Study is to compare the impact on clinical outcomes of 3 different treatment strategies. The first is using medical (drug) therapy alone with standard care. The second strategy is identical medical (drug) therapy as the first group combined with early heart catheterization (within 24 hours) for angiography and if required, intervention. The third treatment strategy is direct admission (within 3 hrs) to the heart catheterization lab for angioplasty.

WEST patients will be enrolled at first medical contact (using emergency medical services, e.g. ambulance) if possible or through Emergency Departments in participating health care facilities.

DETAILED DESCRIPTION:
The principal objective of WEST is to compare the impact on clinical outcomes of the following three treatment groups defined as Group A: optimal pharmacologic therapy (prompt administration of tenecteplase (TNKase) and enoxaparin) at the earliest point of medical contact with usual post MI care; Group B: an identical pharmacological reperfusion strategy followed by an early invasive strategy including timely mechanical intervention, Group C: timely primary percutaneous coronary intervention (PCI), undertaken after enoxaparin and an oral loading dose of clopidogrel.

The secondary objective of WEST is to compare clinical outcomes of patients receiving optimal pharmacologic therapy and a strategy of usual post-MI care, Group A versus protocol-mandated early catheterisation and PCI, Group B.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patients aged >18 years
* Patients with symptoms presumed secondary to STEMI lasting at least 20 minutes and accompanied by ECG evidence >2 mm of ST elevation in 2 or more contiguous precordial leads or in 2 or more limb leads;or > 1mm ST elevation in 2 or more limb leads coupled with >1 mm ST depression in 2 or more contiguous precordial leads such that the total ST deviation is >4 mm; or presumed new left bundle branch block
* Earliest point of care and randomisation must be within 6 hours of onset of symptoms as defined in previous criteria
* Females of child-bearing age, not using a generally accepted method of contraception must have a negative urine pregnancy test
* Written informed consent prior to randomisation of study

Exclusion Criteria:

* PCI expected to commence within < 60 minutes from identification of suitable candidate
* Inability to have angiography/PCI within 3 hrs from randomisation
* Active bleeding or known hemorrhagic diathesis
* Any history of stroke, transient ischemic attack, dementia or structural CNS damage e.g. neoplasm, aneurysm, AV malformation
* Major surgery or trauma within the past 3 months
* Previous Coronary Artery Bypass Graft (CABG)
* Use of abciximab (ReoPro) or other GP IIb/IIIa antagonists within the preceding 7 days
* Any minor head trauma and/or any other trauma occurring after onset of the current myocardial infarction
* Significant hypertension (i.e. SBP > 180 mm HG and/or DBP > 110mm HG) at any time from presentation (earliest point of care) to randomisation
* Current treatment with vitamin K antagonist (warfarin) resulting with an INR > 1.5
* Anticipated difficulty obtaining vascular access
* Prolonged (>10 min) cardiopulmonary resuscitation or cardiogenic shock
* Patients who have participated in an investigational drug study within 7 days prior to randomisation
* Known renal insufficiency (prior creatinine >2.5 mg% for men and >2.0 mg% for women)
* Treatment with standard unfractionated heparin (heparin sodium) >5000 IU or a therapeutic dose of any low molecular weight heparin, within 6 hours prior to randomisation
* Known thrombocytopenia (prior platelet count below 100 000/ul)
* Known sensitivity to TNKase, clopidogrel, heparin, low molecular weight heparin or abciximab
* Pregnancy or lactation, parturition within the previous 30 days
* Any serious concomitant systemic or life limiting disorder that would be incompatible with the trial
* Inability to follow protocol and comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-07

PRIMARY OUTCOMES:
composite of 6 elements defined by: death
recurrent myocardial infarction
heart failure
cardiogenic shock
refractory ischemia
major ventricular arrhythmia

SECONDARY OUTCOMES:
90 and 180 minute ECG ST resolution
QRS determined infarct size at discharge/day 7
CK infarct size determined by area under the curve or peak CK-MB

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. Armstrong, M.D., Study Chair — Canadian VIGOUR Centre
Locations (16):
- Canada (16):
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Misericordia Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Leduc General Hospital, Leduc, Alberta
  - Sturgeon Community Health Care Centre, St. Albert, Alberta
  - Richmond Hospital, Richmond, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Lions Gate Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dartmouth General Hospital, Dartmouth, Nova Scotia
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Cobequid Community Health Centre Emergency Department, Lower Sackville, Nova Scotia
  - Montreal Heart Institute, Montreal, Quebec
  - Pierre Le Gardeur Hospital, Repentigny, Quebec

REFERENCES:
- [Background] Armstrong PW; WEST Steering Committee. A comparison of pharmacologic therapy with/without timely coronary intervention vs. primary percutaneous intervention early after ST-elevation myocardial infarction: the WEST (Which Early ST-elevation myocardial infarction Therapy) study. Eur Heart J. 2006 Jul;27(13):1530-8. doi: 10.1093/eurheartj/ehl088. Epub 2006 Jun 6. PMID 16757491
- [Derived] Westerhout CM, Bonnefoy E, Welsh RC, Steg PG, Boutitie F, Armstrong PW. The influence of time from symptom onset and reperfusion strategy on 1-year survival in ST-elevation myocardial infarction: a pooled analysis of an early fibrinolytic strategy versus primary percutaneous coronary intervention from CAPTIM and WEST. Am Heart J. 2011 Feb;161(2):283-90. doi: 10.1016/j.ahj.2010.10.033. PMID 21315210
- See also: Canadian VIGOUR Centre Homepage — http://www.vigour.ualberta.ca